CLINICAL TRIAL: NCT01759615
Title: A Randomized Clinical Trial on Comparison of Early Versus Late Initiation of Feeding in Preterm Small for Gestation Infants Below 35 Weeks Gestation With Prenatal Absent or Reversal of End Diastolic Flow (AREDF) in Umbilical Artery
Brief Title: Early Versus Late Initiation of Feeding in Preterm Newborns With Prenatal AREDF in Umbilical Artery
Acronym: AREDF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Hardinge Medical College (Other Government)
Collaborators: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sushma Nangia, M.D., Professor, Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: AIIMS/06/AREDF
Record Dates: First submitted 2012-12-23; First posted 2013-01-03 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Time for Achievement of Full Feeds
Keywords: Preterm; SGA; AREDF; Early feeding; Late feeding; Feed intolerence; Necrotizing enterocolitis
MeSH Terms: conditions — Premature Birth; Enterocolitis, Necrotizing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early enteral feeding (Experimental): Early enteral feeding group received minimal enteral feed (MEF) of 8 ml/kg of expressed human milk of the biologic mother for 48 hours followed by regular feeding with feed increments of 20ml/kg/day to reach 150 ml/kg.
  Interventions: Other: Early Enteral feeding
- Late enteral feeding (Active Comparator): Late enteral feeding group was kept NPO for a period of 48 hours followed by minimal enteral feed (MEF) of 8 ml/kg of expressed human milk of the biologic mother for 48 hours and thereafter received regular feeding with feed increments of 20ml/kg/day till full enteral feeds of 150 ml/kg/day were achieved
  Interventions: Other: Late enteral feeding

INTERVENTIONS:
Other: Early Enteral feeding — Feeding with expressed breast milk @ 8ml/kg/day for 48 hrs after randomization at 60+/-12 hrs of life
  Arms: Early enteral feeding
Other: Late enteral feeding — Nil per oral for another 48 hrs after randomization at 60+/-12 hrs of life followed by Feeding with expressed breast milk @ 8ml/kg/day for 48 hrs
  Arms: Late enteral feeding

SUMMARY:
This research is being conducted in preterm newborns with 'in utero' growth restriction due to inadequate blood flow from the mother to the baby. These deprived babies adapt to the not so conducive uterine environment by certain adjustments in blood supply to internal organs thereby permitting as best as possible blood flow to brain heart etc., which are the vital organs and whose adequate functioning is required for survival. In this bargain the gut (intestines) gets poor blood supply and hence its appropriate functioning is jeopardized. In the past such babies (after birth) were not fed for days together which compromised their growth even further. Premature growth restricted' babies are at increased risk of further growth faltering if not fed in time as also to a condition called 'Necrotising enterocolitis' if fed liberally like other healthy neonates, characterized by abdominal distension, blood in stools and inability to feed for much longer duration thereby further affecting growth. This study is evaluating a feeding schedule of early versus late initiation of feeding to arrive at the best time to feed such doubly jeopardized premature growth restricted babies to avert the above mentioned consequences.

No study has been conducted in India to confirm the aforementioned fact and hence this study has been planned. The information learned from this study will help us to feed these small premature as well as growth restricted babies with AREDF better which will go a long way in the care of such preterm growth restricted newborns.

DETAILED DESCRIPTION:
Absence or reversal of end diastolic flow (AREDF) in the umbilical artery is associated with poor outcome. This is further exaggerated by the presence of intrauterine growth retardation and oligohydramnios. Elective premature delivery of such fetuses is common. AREDF leads to circulatory redistribution with decreased blood flow to the lung, intestines, kidneys, skin, and muscle, and blood diverted to the brain, myocardium and adrenals. This reduction in visceral perfusion has been associated with an increased risk of necrotising enterocolitis, cerebral haemorrhage, and neonatal morbidity. Because of concern that feedings may increase the risk of necrotizing enterocolitis, some high-risk infants (most studies on preterm AGA) have received prolonged periods of parenteral nutrition without enteral feedings. Providing trophic feedings (small volume feedings given at the same rate for at least 5 days) during this period of parenteral nutrition was developed as a strategy to enhance feeding tolerance and decrease time to reach full feedings. Whether trophic feedings result in better outcomes than initially withholding feedings or providing progressively increasing feedings can be established only in proper clinical trials.

There are no standard guidelines to feed these preterm SGA infants born to mothers with abnormal antenatal Doppler studies. Furthermore, there are no randomized trials on feeding strategies in this group of neonates and hence we planned to carry out this study on comparison of early versus delayed initiation of feeding in preterm SGA infants with AREDF.

The purpose of this study is to compare the time to reach full enteral feeds, time to regain birth weight etc. in babies who are fed carefully versus those who are not fed for the initial days. It is postulated that early gut priming may stimulate the gut to secrete certain trophic and growth factors which may make it better able to tolerate enteral feeds improving the overall growth and also reducing chances of infection.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm neonates below 35 weeks gestation born at the study center(s)
2. Small for gestational age (SGA) ie weight < 10th centile for gestation
3. Absent or reverse end diastolic flow (AREDF) in umbilical artery'

Exclusion Criteria:

1. Babies with major congenital malformations.
2. Babies with severe asphyxia as defined by apgar score <4 at 5 min of life with cord/within one hour of life pH< 7.0.
3. Shock requiring pressor support at the time of randomization.
4. Babies born with gastrointestinal surgical conditions precluding enteral feeding.
5. Babies with abdominal distension, bilious or hemorrhagic aspirates or recurrent vomiting at the time of randomization.
6. Refusal to obtain consent.
7. Gestation below 26 weeks.
8. Hydrops fetalis.

Min Age: 60 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-04; Primary Completion 2007-02 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Time taken to achieve full feeds | in days upto six weeks
  First day of the three days when full enteral feeding of 150 ml/kg has been achieved and sustained as recorded from the nursing chart of the infant.

SECONDARY OUTCOMES:
Days to regain birth weight | in days upto six weeks
  After the initial fall in weight the first day when birth weight is regained or crossed and the value remains above the birth weight for subsequent 2 days will be recorded as day of life birth weight has been regained.
Feed intolerance | till achievement of full feeds
  Feed intolerance was measured as number of episodes of any of the following symptoms per infant till he/she reached full feeds of 150ml/kg and sustained it for 2 days.
  * bilious or hemorrhagic aspirates( irrespective of the volume),
  * vomiting ( >2 times in 12 hours duration) and
  * clear or milky aspirate >50% of the previous feed volume necessitating feed stoppage for 24 hours
duration of stay | in days upto twelve weeks
  This was taken to be the interval between birth and the day the newborn was discharged home.

CONTACTS AND LOCATIONS:
Overall Officials: Sushma Nangia, MD, DM, Principal Investigator — All India Institute of Medical Sciences